CLINICAL TRIAL: NCT01085396
Title: Optical Spectroscopy for Non-invasive Diagnosis of Melanoma and Assessment of Impact of UV Exposure on Skin
Brief Title: Use of Fiber-optic Probe for Non-invasive Diagnosis of Melanoma and Assessment of Impact of Ultraviolet (UV) Exposure on Skin
Status: Terminated | Type: Observational
Why Stopped: Ran out of funding
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Yang Liu, PhD, Principal Investigator, University of Pittsburgh
Other Study IDs: UPCI 09-077
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2014-05

CONDITIONS: Melanoma
Keywords: Fiber Optic; Melanoma; UV Exposure
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A pigmented lesion is removed as part of the subjects routine care when it is felt to be suspicious for severe atypica or early malignancy, and sometimes because the patient desires removal of lesions for cosmetic reasons, or because the lesion is irritated or located in a zone of traum.
  For this research study, samples of the tumor tissue from these clinical care biopsies will be studied.
  Researchers will look at markers and search for additional characteristics that may help them better understand Melanoma. This will be optional to subjects. If subjects do not agree to have their tissue kept for future research purposes they can still participate in the rest of this study.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is designed to collect information about melanoma using a research probe, a device placed only on the skin. This study will investigate whether using the probe to examine skin lesions could improve the accuracy of identification pre-cancerous melanoma lesions or to predict the risk melanoma in the skin of subjects. Ultimately, we would see this technique used routinely as a non-invasive device during subjects' skin examination to aid dermatologists to identify pre-cancerous (melanoma) lesions without taking tissue samples of the skin. Alternatively, this technique would, in the future, also be used to screen patients at risk for melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Male and female above 18 years of age;
* Subjects who are planned to undergo skin examinations with and without atypical nevi, with and without personal or family history of melanoma and potentially with pigmented lesions to be removed for medical care or cosmetic purposes.

Exclusion Criteria:

* Individuals whose pathology cannot be obtained or retrieved.
* Inability to provide informed consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. normal volunteers
  2. patients without personal and family history of melanoma
  3. patients with personal or family history of melanoma who are followed in the UPCI Melanoma Program with either atypical nevi or without atypical nevi.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2010-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Investigate the ability of the fiber-optic probe to identify lesions of melanoma and severe/high-grade dysplasia | 3 years
  To correct for skin color effect and heterogeneity, the readings of the pigmented lesion will be normalized by the readings taken from the corresponding normal skin around the lesion.

SECONDARY OUTCOMES:
To test whether the fiber-optic probe can discriminate the severe/high-grade dysplasia from the mild and moderate dysplastic nevi; | 3 years
To test whether the fiber-optic probe readings are different among tissues with different degree of sun exposure | 3 years
To test whether the fiber-optic probe readings are different between the most and the least suspicious lesions | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yang Liu, PhD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - UPMC Presbyterian Dept. of Dermatology, Pittsburgh, Pennsylvania
  - UPCI - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Shadyside Place - Dermatology Unit, Pittsburgh, Pennsylvania